CLINICAL TRIAL: NCT04232930
Title: The Use of Music in Reducing Pain During Outpatient Hysteroscopy: Prospective Randomized Trial
Brief Title: The Use of Music in Reducing Pain During Outpatient Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Principal Investigator, Law Ho Ying, Resident, Department of Obstetrics and Gynaecology, Pamela Youde Nethersole Eastern Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HKECREC-2019-034
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Hysteroscopy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Prospective randomized trial
Masking Description: This is not a blinded study as both the participant and the care provider will be able to listen to the music if the subject is assigned into the music group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music group (Active Comparator): In the music group, music that chosen by the participant will be played through a speaker by the nursing staff during outpatient hysteroscopy. Music will be played through a speaker instead of headphone in order to maintain a good communication and interaction between the participant and the doctor.
  Interventions: Other: Music
- Non-music group (No Intervention): Participants in the non-music group will undergo outpatient hysteroscopy in the same setting and standard procedure without listening to any music.

INTERVENTIONS:
Other: Music — Four types of music will be provided, including pop, classical, jazz or spa music which are prepared by the study team. They contain instrumental songs only without vocal.
  Arms: Music group

SUMMARY:
The aim of this study is to demonstrate the value of music in outpatient hysteroscopy on patients' level of pain and satisfaction. This may have a role in our daily practice in providing a better patient care in outpatient hysteroscopy.

DETAILED DESCRIPTION:
Outpatient hysteroscopy is nowadays a commonly used procedure in Gynaecology in order to evaluate the uterine cavity and to diagnose different intrauterine diseases. It is a safe, convenient and cost-effective procedure in aiding the management of abnormal uterine bleeding. However, outpatient hysteroscopy can be associated with significant pain which would have impact on the woman's satisfaction and pain is one of the most common reasons for failure of the procedure.

Listening to music could be an easy and non-invasive way to reduce pain. A meta-analysis conducted on the effects of music on pain revealed that music interventions had statistically significant effects in decreasing pain on 0-10 pain scales. Researches on this topic in gynaecological office procedures, however, showed variation in the results. Some showed no positive effect of music on patient's level of pain, anxiety or satisfaction of patient or doctor for office hysteroscopy and colposcopy. On the other hand, some studies showed a positive effect of the use of music with a reduction of pain and anxiety during office hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* indication for hysteroscopy (abnormal uterine bleeding, abnormal findings on ultrasound, and infertility)
* signed informed consent
* ability to read Chinese or English.

Exclusion Criteria:

* hearing impairment
* known anatomical abnormalities which would make performing the procedure more difficult
* use of premedication for cervical ripening

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Intensity of pain | Anticipated pain before hysteroscopy
  Pain measured using visual analog scale (VAS) on a 0-10 scale, with 0 indicating "no pain" and 10 indicating "worst pain possible".
Intensity of pain | Actual pain experienced during hysteroscopy
  Pain measured using visual analog scale (VAS) on a 0-10 scale, with 0 indicating "no pain" and 10 indicating "worst pain possible".

SECONDARY OUTCOMES:
Systolic blood pressure | Systolic blood pressure before hysteroscopy
  Systolic blood pressure
Systolic blood pressure | Systolic blood pressure during hysteroscopy
  Systolic blood pressure
Diastolic blood pressure | Diastolic blood pressure before hysteroscopy
  Diastolic blood pressure
Diastolic blood pressure | Diastolic blood pressure during hysteroscopy
  Diastolic blood pressure
Heart rate | Heart rate before hysteroscopy
  Heart rate
Heart rate | Heart rate during hysteroscopy
  Heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Ho Ying Law, Principal Investigator — Pamela Youde Nethersole Eastern Hospital
Locations (1):
- Pamela Youde Nethersole Eastern Hospital, Hong Kong, HongKong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The following individual participant data will be shared:
  * Background characteristics including age, body mass index, occupation, religion, education, marital status, parity and number of vaginal deliveries and history of hysteroscopic surgery
  * Details of the outpatient hysteroscopy including time, procedure and level of performing surgeon
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The personal data will be kept for 3 years after the study. All the personal data will be discarded and destroyed after the storage period.
Access Criteria: When a third party is interested to reanalyze study data or to combine data from multiple studies.

REFERENCES:
- [Background] Morgan M, Dodds W, Wolfe C, Raju S. Women's views and experiences of outpatient hysteroscopy: implications for a patient-centered service. Nurs Health Sci. 2004 Dec;6(4):315-20. doi: 10.1111/j.1442-2018.2004.00202.x. PMID 15507052
- [Background] Amer-Cuenca JJ, Marin-Buck A, Vitale SG, La Rosa VL, Caruso S, Cianci A, Lison JF. Non-pharmacological pain control in outpatient hysteroscopies. Minim Invasive Ther Allied Technol. 2020 Feb;29(1):10-19. doi: 10.1080/13645706.2019.1576054. Epub 2019 Feb 22. PMID 30794005
- [Background] Mak N, Reinders IMA, Slockers SA, Westen EHMN, Maas JWM, Bongers MY. The effect of music in gynaecological office procedures on pain, anxiety and satisfaction: a randomized controlled trial. Gynecol Surg. 2017;14(1):14. doi: 10.1186/s10397-017-1016-2. Epub 2017 Aug 9. PMID 28890676
- [Background] Angioli R, De Cicco Nardone C, Plotti F, Cafa EV, Dugo N, Damiani P, Ricciardi R, Linciano F, Terranova C. Use of music to reduce anxiety during office hysteroscopy: prospective randomized trial. J Minim Invasive Gynecol. 2014 May-Jun;21(3):454-9. doi: 10.1016/j.jmig.2013.07.020. Epub 2013 Aug 17. PMID 23962572
- [Background] Chan YM, Lee PW, Ng TY, Ngan HY, Wong LC. The use of music to reduce anxiety for patients undergoing colposcopy: a randomized trial. Gynecol Oncol. 2003 Oct;91(1):213-7. doi: 10.1016/s0090-8258(03)00412-8. PMID 14529684
- [Background] Lee JH. The Effects of Music on Pain: A Meta-Analysis. J Music Ther. 2016 Winter;53(4):430-477. doi: 10.1093/jmt/thw012. Epub 2016 Oct 19. PMID 27760797
- See also: Best Practice in Outpatient Hysteroscopy — https://www.rcog.org.uk/globalassets/documents/guidelines/gtg59hysteroscopy.pdf

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT04232930/Prot_SAP_ICF_002.pdf